CLINICAL TRIAL: NCT01409031
Title: Phase II Trial of Sildenafil in Newborns With Persistent Pulmonary Hypertension
Brief Title: Study of Sildenafil to Treat Newborns With Persistent Pulmonary Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial was terminated early due to lack of recruitment.
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); State University of New York at Buffalo (Other); Vanderbilt University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Utah (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-1211; 1U01HL102235 (NIH)
Record Dates: First submitted 2011-07-15; First posted 2011-08-03 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Persistent Pulmonary Hypertension; Respiratory Failure
Keywords: newborns; respiratory failure; pulmonary hypertension; treatment
MeSH Terms: conditions — Respiratory Insufficiency; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous Sildenafil (Experimental)
  Interventions: Drug: Intravenous Sildenafil
- Placebo (Placebo Comparator): 0.4 mg/kg bolus, followed by a continuous infusion of 1.6 mg/kg/day or an equivalent volume of placebo (D5W); infusion will be initiated as a bolus over 3 hours, followed by a controlled continuous infusion for up to 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intravenous Sildenafil — 0.4 mg/kg bolus, followed by a continuous infusion of 1.6 mg/kg/day or an equivalent volume of placebo (D5W); infusion will be initiated as a bolus over 3 hours, followed by a controlled continuous infusion for up to 7 days.
  Other Names: Revatio
  Arms: Intravenous Sildenafil
Other: Placebo — An equivalent volume of placebo (D5W)infusion will be initiated as a bolus over 3 hours, followed by a controlled continuous infusion for up to 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intravenous sildenafil reduces pulmonary artery pressure and improves oxygenation in near-term and term infants with persistent pulmonary hypertension.

DETAILED DESCRIPTION:
Term infants with respiratory failure and persistent pulmonary hypertension (PPHN) are among the most critically ill infants in the NICU, with significant mortality and morbidity reported even for infants with moderate disease. Currently, management is largely supportive, and includes oxygen, mechanical ventilation (conventional or high frequency ventilation), and exogenous surfactant therapy. Inhaled nitric oxide (iNO) is a pulmonary vasodilator that was approved for the treatment of hypoxic respiratory failure (HRF) and PPHN of the newborn in 1999 based on clinical trials showing a reduction in the need for rescue treatment with extracorporeal membrane oxygenation (ECMO).

One promising therapy to decrease pulmonary arterial pressure and improve oxygenation is sildenafil. Sildenafil is a cGMP-specific phosphodiesterase inhibitor that causes relatively selective pulmonary vasodilation. The use of intravenous (IV) sildenafil was recently FDA approved for use in adults in PPHN. A pilot trial studying dose response and pharmacokinetics in 36 term newborns with PPHN found that IV sildenafil was well tolerated and has the potential to induce marked improvements in oxygenation. The data from this pilot trial provided background to support the dosing regimen for this Phase II trial. We hypothesize that IV sildenafil will acutely reduce pulmonary artery pressure and improve oxygenation in near-term and term infants with PPHN, thus reducing the need for rescue therapy iNO and/or ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from legally acceptable guardian
* PPHN or hypoxemic respiratory failure associated with:

  * Idiopathic PPHN
  * Meconium aspiration syndrome
  * Respiratory distress syndrome
  * Sepsis
  * Pneumonia
* Greater than or equal to 35 weeks gestation
* Age at enrollment less than 72 hours
* Moderate hypoxemic respiratory failure, with 12<OI<35 (oxygenation index, calculated as FiO2 * mean airway pressure * 100 / postductal PaO2)
* Absence of structural heart disease (except patent ductus arteriosus, atrial septal defect <1cm, or muscular ventricular septal defect < 2mm)
* Absence of lethal congenital anomaly
* Not participating in another concurrent experimental study

Exclusion Criteria:

* Prior or immediate need for iNO or ECMO
* Profound hypoxemia: qualifying PaO2 <30 mmHg, from a blood gas drawn within 30 minutes of starting study drug infusion.
* Hypotension: Mean arterial pressure <35 mmHg
* Congenital heart disease, except patent ductus arteriosus, atrial septal defect <1cm, or muscular ventricular septal defect <2mm
* Congenital diaphragmatic hernia or lung hypoplasia syndromes, diagnosed on the basis of prolonged oligohydramnios
* Active seizures
* Apgar score of <3 at 5 minutes
* Bleeding diathesis
* Receipt of any other experimental drug or device
* Receipt of any prohibited concurrent medication:

  * Potent cytochrome P450 3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole and protease inhibitors)
  * Endothelin antagonists (e.g. Tracleer/bosentan)
  * Intravenous nitrates or nitric oxide donors
* Known hereditary degenerative retinal disorders such as retinitis pigmentosa.
* In the opinion of the investigator, a subject who is not likely to complete the study or would be considered inappropriate for the study, for any reason.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kinsella, MD, Principal Investigator — University of Colorado, Denver
Locations (7):
- United States (7):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Anne and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Women's & Children's Hospital of Buffalo SUNY, Buffalo, New York
  - Vanderbilt University, Nashville, Tennessee
  - Primary Children's Medical Center, Utah, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was terminated early due to lack of recruitment.
Period: Overall Study
Arm/Group | Intravenous Sildenafil | Placebo
Started | 1 | 2
Completed | 0 | 2
Not Completed | 1 | 0
Not completed — transferred to other hosp | 1 | 0

BASELINE CHARACTERISTICS:
Population: Newborns meeting entry criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Sildenafil | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Customized [Number; unit: participants] — Age of Newborns in days
  participants
    <=1 days old | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Oxygenation
Time Frame: From baseline values at 4 and 24 hours
Population: This trial was terminated early due to lack of recruitment. No participants completed the study. Data required to assess this outcome measure was not collected.
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Receipt of Standard Therapy at Any Point During the 7-day Treatment Period
Description: Receipt of standard therapy (inhaled nitric oxide [iNO] and/or extracorporeal membrane oxygenation [ECMO]) at any point during the 7-day treatment period
Time Frame: 7-day treatment period
Population: as for outcome 1
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Pulmonary Arterial Pressure
Description: Change in pulmonary arterial pressure as calculated by echocardiography
Time Frame: Baseline and 4 hours post study drug administration
Population: as for outcome 1
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Supplemental O2
Time Frame: Participants will be on supplemental O2 an average of 2 weeks
Population: as for outcome 1
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Age at Hospital Discharge
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Population: as for outcome 1
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: Participants will be on mechanical ventilation an average of 1 week
Population: as for outcome 1
Arm/Group | Intravenous Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Sildenafil (N=1) | Placebo (N=2)
PaO2 < 40 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Given that this trial was stopped with only 3 patients randomized, the results are little more than anecdote except that the participants were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No